CLINICAL TRIAL: NCT01107964
Title: Oral Omega-3 Fatty Acids in the Treatment of Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: The American Society of Cataract and Refractive Surgery Foundation (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, David Liang, Physician, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33794
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; Recent Diagnosis of Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3-acid ethyl esters (Active Comparator)
  Interventions: Drug: Oral Omega-3-acid ethyl esters
- Corn oil capsule (Placebo Comparator)
  Interventions: Drug: Placebo corn oil capsule

INTERVENTIONS:
Drug: Oral Omega-3-acid ethyl esters — 1 gram capsule by mouth four times daily for 45 days
  Arms: Omega-3-acid ethyl esters
Drug: Placebo corn oil capsule — 1 gram by mouth 4 times daily for 45 days
  Arms: Corn oil capsule

SUMMARY:
The investigators hypothesize that oral omega-3-acid ethyl esters (Lovaza, GlaxoSmithKline, Research Triangle Park, NC) will decrease dry-eye related symptoms as well as clinical markers associated with dry eye disease (Schirmer-1 test values, positive vital staining with lissamine green, and fluorescein tear break-up time) when compared to administration of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Typical symptoms of dry eye (photophobia, burning, foreign body sensation, blurred vision improved with blinking)
* Schirmer Test < 8 mm/5 minutes
* Fluorescein tear break-up time < 8 seconds
* No current use of dry eye treatment (except artificial lubrication)
* Signature on consent form

Exclusion Criteria:

* Infectious keratoconjunctivitis or inflammatory disease unrelated to dry eye
* Eyelid or eyelash abnormalities
* Alteration of the nasolacrimal apparatus
* Treatment with drugs affecting tearing
* Concomitant ocular therapies
* Topical ophthalmic steroids taken during the 4 weeks before the study
* Pregnant/breast-feeding women
* History of liver disease
* History of fish and/or shellfish allergy or hypersensitivity
* History of corn allergy or hypersensitivity
* Treatment with systemic anticoagulation therapy
* Patients with bleeding disorders or those receiving anticoagulation (e.g., warfarin, enoxaparin, dipyridamole, clopidogrel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Liang, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Eye Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule
Started | 13 | 14
Completed | 12 | 13
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [44.5 to 65] | 60 [55 to 67] | 58 [49.5 to 67.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Ocular Surface Disease Index Score at Day 45
Description: The Ocular Surface Disease Index Score is a validated, scored questionnaire that measures subjective symptoms of dry eye. Possible scores range from 0 (no symptoms of dry eye) to 100 (severest symptoms of dry eye). Change = (Day 45 score - Baseline score)
Time Frame: Baseline and Day 45
Population: Throughout the study, we evaluated the worse eye of each patient, defined as the eye with the the higher Lissamine Green Staining Score or the eye with the lower Schirmer-1 Test Value in the event of equality.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule
Number analyzed (Participants) | 12 | 13
Number analyzed (eyes) | 12 | 13
units on a scale | -28.4 [-36.4 to -11.8] | -5.8 [-39.6 to 1.3]
Statistical Analysis 1: Comparison: Omega-3-acid Ethyl Esters vs Corn Oil Capsule; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline of Schirmer-1 Test Value at Day 45
Description: Schirmer-1 Test Value is a measurement of tear production. The amount of tears are measured in total millimeters after 5 minutes has elapsed. Low levels of tear production are associated with dry eye. Change = (Day 45 value - Baseline value).
Time Frame: Baseline and Day 45
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: millimeters
Units Other Than Participants: eyes
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule
Number analyzed (Participants) | 12 | 13
Number analyzed (eyes) | 12 | 13
millimeters | -2.5 [-3.0 to 1.0] | 1.0 [-4.0 to 4.0]
Statistical Analysis 1: Comparison: Omega-3-acid Ethyl Esters vs Corn Oil Capsule; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline of Lissamine Green Staining Score at Day 45
Description: Lissamine Green Staining Score is a measure of ocular surface irregularity secondary to dry eye. Possible scores range from 0 (no ocular surface irregularity secondary to dry eye) to 9 (severe ocular surface irregularity secondary to dry eye). Change = (Day 45 score - Baseline score)
Time Frame: Baseline and Day 45
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule
Number analyzed (Participants) | 12 | 13
Number analyzed (eyes) | 12 | 13
units on a scale | 1.0 [-1.5 to 1.0] | -1.0 [-2.0 to 0]
Statistical Analysis 1: Comparison: Omega-3-acid Ethyl Esters vs Corn Oil Capsule; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline of Fluorescein Tear Break-Up Time (Seconds) at Day 45
Description: Fluorescein Tear Break-Up Time is a measurement in seconds of tear film stability. The shorter the Fluorescein Tear Break-Up Time, the lower the tear film stability.
  Lower tear film stability is associated with dry eye. Change = (Day 45 value - Baseline value).
Time Frame: Baseline and Day 45
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: time in seconds
Units Other Than Participants: eyes
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule
Number analyzed (Participants) | 12 | 13
Number analyzed (eyes) | 12 | 13
time in seconds | 1.7 [0.3 to 3.8] | 0.3 [-0.7 to 4.3]
Statistical Analysis 1: Comparison: Omega-3-acid Ethyl Esters vs Corn Oil Capsule; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire duration of the 45 day trial.
Arm/Group | Omega-3-acid Ethyl Esters | Corn Oil Capsule
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 2/13 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3-acid Ethyl Esters (N=13) | Corn Oil Capsule (N=14)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes